CLINICAL TRIAL: NCT04015934
Title: Predictive Factors Identification of Long-term Outcome in Multifocal Motor Neuropathy (MMN) Treated With Intravenous Immunoglobulin (IVIG)
Brief Title: Predictive Factors of Long Term Outcome in MMN
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Régional Metz-Thionville (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: NMMBC
Record Dates: First submitted 2019-05-31; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-05

CONDITIONS: MMN
Keywords: predictive factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cornerstone treatment for multifocal motor neuropathy (MMN), a rare and disabling dysimmune neuropathy, is intravenous immunoglobulin (IVIg). The aim of this study is to identify prognostic factors of poor outcome.

Data were retrospectively collected from MNN patients in three French centers. Patients were divided into two groups: a good outcome group and a poor outcome group. Demographic, clinical, biological and nerve conduction study features of MMN patients were analyzed. Identification of prognostic factors in MMN could help develop personalized treatment.

DETAILED DESCRIPTION:
The cornerstone treatment for multifocal motor neuropathy (MMN), a rare and disabling dysimmune neuropathy, is intravenous immunoglobulin (IVIg). However, 10% of patients progress despite treatment. The aim of this study is to identify prognostic factors of poor outcome.

Data were retrospectively collected from MNN patients in three French centers. Patients were divided into two groups: a good outcome group (patients in remission without IVIg or with spaced IVIg courses), and a poor outcome group (patients dependent on continuous IVIg treatment or deteriorating despite IVIg). Investigators searched predictive factors of long-term outcome in MMN. They studied demographic, clinical, biological and nerve conduction study features of MMN patients.Identification of prognostic factors in MMN could help develop personalized treatment by selecting patients eligible for immunosuppressive drugs before IVIg dependence or progression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MNN following the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) Guideline criteria 2010

Exclusion Criteria:

* missing data
* clinical progression features suggested another inflammatory neuropathy,
* immunosuppressive agents for another pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MMN patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Presence of deteriorating or strongly dependant IVIg NMM | inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: No